CLINICAL TRIAL: NCT00002723
Title: A PHASE III STUDY OF THREE DIFFERENT DOSES OF SURAMIN (NSC #34936) ADMINISTERED WITH A FIXED DOSING SCHEDULE IN PATIENTS WITH ADVANCED PROSTATE CANCER
Brief Title: Low, Intermediate, or High Dose Suramin in Treating Patients With Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: SWOG Cancer Research Network (Network); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02788; U10CA031946 (NIH); CALGB-9480; E-C9480; SWOG-9452; INT-0159; CDR0000064583 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-10-22 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Suramin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose suramin (Experimental): Low dose suramin
  Interventions: Drug: suramin
- Intermediate dose suramin (Experimental): Intermediate dose suramin
  Interventions: Drug: suramin
- High dose suramin (Experimental): High dose suramin
  Interventions: Drug: Suramin

INTERVENTIONS:
Drug: suramin — 3.192g/square meter total dose given decreasing concentrations in 250 cc normal saline IV over 1 hour on days 1,2,8,9,29,30,36,37,57,58,64,and 65.
  Other Names: NSC #34936
  Arms: Low dose suramin
Drug: suramin — 5.320 g/square meter total dose given in decreasing concentrations in 250 cc normal saline via IV over 1 hour on days 1,2,8,9,29,30,36,37,57,58,64,and 65
  Other Names: NSC #34936
  Arms: Intermediate dose suramin
Drug: Suramin — 7.661 g/square meter toal dose given in decreasing concentrations in 250 cc normal saline IV over 1 hour on days 1,2,8,9,29,30,36,37,5,58,64,and 65.
  Other Names: NSC #34936
  Arms: High dose suramin

SUMMARY:
Randomized phase III trial to compare the effectiveness of low, intermediate, and high dose suramin in treating men with stage IV prostate cancer that is refractory to hormone therapy. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which regimen of suramin is more effective for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the response in patients with advanced hormone-refractory adenocarcinoma of the prostate treated with low- vs intermediate- vs high-dose suramin.

II. Compare the toxic effects of these regimens in these patients. III. Compare the overall and failure-free survival of patients treated with these regimens.

IV. Compare the duration of complete and partial responses in patients treated with these regimens.

V. Determine the population pharmacokinetics of these regimens and correlate these parameters with the toxicity of these regimens and response rate in these patients.

VI. Compare the quality of life of patients treated with these regimens. VII. Determine the relationship of absolute and relative decrease in PSA and rate of PSA decrease with the likelihood and duration of response in patients treated with these regimens.

VIII. Determine whether a change in fibroblast growth factor levels in patients treated with suramin can be associated with the pharmacokinetics of suramin or the likelihood of clinical response in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease site (bone only vs soft tissue), CALGB/Zubrod performance status (0 or 1 vs 2), number of prior hormonal therapies (1 or 2 vs 3), and participating center. Patients are randomized to 1 of 3 treatment arms.

Arm I: Patients receive low-dose suramin IV over 1 hour on days 1, 2, 8, 9, 29, 30, 36, 37, 57, 58, 64, and 65 in the absence of disease progression or unacceptable toxicity.

Arm II: Patients receive intermediate-dose suramin as in arm I.

Arm III: Patients receive high-dose suramin as in arm I. Patients with new progression after partial or complete response may receive additional courses, at the discretion of the study chairperson, beginning at least 12 weeks after completion of the first course and continuing in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed.

Patients are followed every 4 weeks until disease progression and then periodically for new primary cancer(s) and survival.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven adenocarcinoma of the prostate with progressive metastatic or progressive regional nodal disease

  * PSA evidence of progression defined as at least 50% increase over baseline on at least 2 measurements at least 2 weeks apart
* Measurable disease preferred but not required

  * Bone scan abnormalities acceptable provided PSA at least 10 ng/mL
  * No minimum PSA value required if measurable disease present
* Progression after or during an adequate trial of hormonal therapy
* No more than 3 prior hormonal interventions for progressive disease

  * One prior hormonal intervention is defined by any of the following:

    * Concurrent testicular and adrenal androgen ablation (e.g., leuprolide, goserelin, orchiectomy, or diethylstilbestrol (DES) plus flutamide, bicalutamide, nilutamide, megestrol, or other antiandrogen)
    * Initial LHRH agonist followed by orchiectomy provided no progression prior to orchiectomy
    * Prior intermittent androgen deprivation on protocol SWOG-9346
    * Corticosteroids for metastatic disease or in conjunction with aminoglutethimide or ketoconazole
  * Two prior hormonal interventions are defined by the following:

    * Antiandrogen given for disease progression more than 3 months after initial hormonal therapy
* Prior neoadjuvant or adjuvant deprivation for treatment of nonmetastatic disease not considered a prior hormonal intervention
* Antiandrogen withdrawal not considered a separate hormonal intervention

  * At least 4 weeks since antiandrogen withdrawal or megestrol withdrawal
  * Failure to respond to (i.e., no decrease in PSA at 2 and 4 weeks) or progression after a transient response to antiandrogen withdrawal or megestrol withdrawal required
* Primary testicular androgen suppression (e.g., LHRH agonist or DES) continues during study
* No brain metastases or other CNS disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* CALGB 0-2 OR
* Zubrod 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm3
* Absolute neutrophil count at least 1,200/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 9 g/dL
* Fibrinogen at least 200 mg/dL
* No prior hemorrhagic or thrombotic disorders

Hepatic:

* Bilirubin normal
* AST/ALT no greater than 2.5 times normal
* Prothrombin time, partial thromboplastin time, and thrombin time normal

Renal:

* Creatinine clearance at least 70 mL/min

Other:

* No primary muscle disease
* No active, uncontrolled bacterial, viral, or fungal infection
* No grade 1 or worse peripheral neuropathy
* No underlying medical condition that would preclude study
* No other serious medical illness that limits survival to less than 3 months
* No psychiatric condition that would preclude informed consent
* No other malignancy within the past 5 years except inactive nonmelanomatous skin cancer or adequately treated stage I or II cancer in remission

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy for metastatic disease

Chemotherapy:

* No prior chemotherapy (including estramustine) for metastatic disease

Endocrine therapy:

* No concurrent megestrol or other hormonal agents
* No concurrent systemic or inhaled corticosteroids (intranasal and topical steroids allowed)

Radiotherapy:

* At least 4 weeks since prior radiotherapy (8 weeks for strontium therapy)

Other:

* No prior experimental therapy for metastatic disease
* No concurrent heparin, warfarin, or aspirin

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 1996-01; Primary Completion 2002-08 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Response | Week 12 and then monthly
  PSA levels
Response | Week 12 and every 12 weeks thereafter
  Radiographic evaluation

SECONDARY OUTCOMES:
Toxicity | pre-study, day 1, then every 2 weeks during treatment and every 8 weeks during follow up
Survival | post treatment until patient expires
Quality of Life | pre-study, 2 weeks post treatment, and every 12 weeks in follow up

CONTACTS AND LOCATIONS:
Overall Officials: Eric J. Small, MD, Study Chair — University of California, San Francisco; Daniel P. Petrylak, MD, Study Chair — Herbert Irving Comprehensive Cancer Center; George Wilding, MD, Study Chair — University of Wisconsin, Madison
Locations (27):
- United States (26):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Pretoria Academic Hospitals, Pretoria, South Africa

REFERENCES:
- [Background] Halabi S, Vogelzang NJ, Kornblith AB, Ou SS, Kantoff PW, Dawson NA, Small EJ. Pain predicts overall survival in men with metastatic castration-refractory prostate cancer. J Clin Oncol. 2008 May 20;26(15):2544-9. doi: 10.1200/JCO.2007.15.0367. PMID 18487572
- [Background] D'Amico AV, Halabi S, Vogelzang NJ, et al.: A reduction in the rate of PSA rise following chemotherapy in patients with metastatic hormone refractory prostate cancer (HRPC) predicts survival: results of a pooled analysis of CALGB HRPC trials. [Abstract] J Clin Oncol 22 (Suppl 14): A-4506, 383s, 2004.
- [Background] Halabi S, Small EJ, Kantoff PW, Kattan MW, Kaplan EB, Dawson NA, Levine EG, Blumenstein BA, Vogelzang NJ. Prognostic model for predicting survival in men with hormone-refractory metastatic prostate cancer. J Clin Oncol. 2003 Apr 1;21(7):1232-7. doi: 10.1200/JCO.2003.06.100. PMID 12663709
- [Background] Gilligan TD, Halabi S, Kantoff PW, et al.: African-American race is associated with longer survival in patients with metastatic hormone-refractory prostate cancer (HRCaP) in four randomized phase III Cancer and Leukemia Group B (CALGB) trials. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-725, 2002.
- [Result] George DJ, Halabi S, Shepard TF, Sanford B, Vogelzang NJ, Small EJ, Kantoff PW. The prognostic significance of plasma interleukin-6 levels in patients with metastatic hormone-refractory prostate cancer: results from cancer and leukemia group B 9480. Clin Cancer Res. 2005 Mar 1;11(5):1815-20. doi: 10.1158/1078-0432.CCR-04-1560. PMID 15756004
- [Result] Taplin ME, George DJ, Halabi S, Sanford B, Febbo PG, Hennessy KT, Mihos CG, Vogelzang NJ, Small EJ, Kantoff PW. Prognostic significance of plasma chromogranin a levels in patients with hormone-refractory prostate cancer treated in Cancer and Leukemia Group B 9480 study. Urology. 2005 Aug;66(2):386-91. doi: 10.1016/j.urology.2005.03.040. PMID 16098367
- [Result] Ahles TA, Herndon JE 2nd, Small EJ, Vogelzang NJ, Kornblith AB, Ratain MJ, Stadler W, Palchak D, Marshall ME, Wilding G, Petrylak D, Holland JC; Cancer and Leukemia Group B. Quality of life impact of three different doses of suramin in patients with metastatic hormone-refractory prostate carcinoma: results of Intergroup O159/Cancer and Leukemia Group B 9480. Cancer. 2004 Nov 15;101(10):2202-8. doi: 10.1002/cncr.20655. PMID 15484217
- [Result] Taplin ME, George DJ, Halabi S, et al.: Prognostic significance of plasma chromogranin A levels in hormone-refractory prostate cancer patients treated on Cancer and Leukemia Group B (CALGB) 9480. [Abstract] J Clin Oncol 22 (Suppl 14): A-4557, 396s, 2004.
- [Result] Small EJ, Halabi S, Ratain MJ, Rosner G, Stadler W, Palchak D, Marshall E, Rago R, Hars V, Wilding G, Petrylak D, Vogelzang NJ. Randomized study of three different doses of suramin administered with a fixed dosing schedule in patients with advanced prostate cancer: results of intergroup 0159, cancer and leukemia group B 9480. J Clin Oncol. 2002 Aug 15;20(16):3369-75. doi: 10.1200/JCO.2002.10.022. PMID 12177096
- [Result] Bok RA, Halabi S, Fei DT, Rodriquez CR, Hayes DF, Vogelzang NJ, Kantoff P, Shuman MA, Small EJ. Vascular endothelial growth factor and basic fibroblast growth factor urine levels as predictors of outcome in hormone-refractory prostate cancer patients: a cancer and leukemia group B study. Cancer Res. 2001 Mar 15;61(6):2533-6. PMID 11289126
- [Result] George DJ, Halabi S, Shepard TF, Vogelzang NJ, Hayes DF, Small EJ, Kantoff PW; Cancer and Leukemia Group B 9480. Prognostic significance of plasma vascular endothelial growth factor levels in patients with hormone-refractory prostate cancer treated on Cancer and Leukemia Group B 9480. Clin Cancer Res. 2001 Jul;7(7):1932-6. PMID 11448906
- [Result] Bok R, Halabi S, Shaal M, et al.: VEGF and basic FGF urine levels as predictors of response to therapy with suramin in CALGB 9480, a phase III study of hormone refractory prostate cancer (HRPC) patients. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A1367, 2000.
- [Result] Halabi S, Small EJ, Ansari RH, et al.: Results of CALGB 9480, a phase III trial of 3 different doses of suramin for the treatment of horomone refractory prostate cancer (HRPC). [Abstract] Proceedings of the American Society of Clinical Oncology 19: A1291, 2000.
- [Result] Kantoff P, Halabi S, Farmer D, et al.: RT-PCR for prostate specific antigen (PSA) in peripheral blood (PB) predicts survival duration in patients with hormone refractory prostate cancer (HRPC): a CALBG study. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A1323, 2000.
- [Result] Vogelzang N, Small E, Halabi R, et al.: A phase III trial of 3 different doses of suramin (SUR) in metastatic hormone refractory prostate cancer (HRPC): safety profile of CALGB 9480. [Abstract] Proceedings of the American Society of Clinical Oncology 17: A1339, 347a, 1998.